CLINICAL TRIAL: NCT01995760
Title: The Most Appropriate Parameter Correlates With Clinical Effectiveness of Vancomycin: Trough Drug Concentration or Area Under Curve (AUC)/Minimum Inhibitory Concentration (MIC)?
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201310037RINA
Record Dates: First submitted 2013-11-10; First posted 2013-11-27 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Methicillin-resistant Staphylococcus Aureus Septicemia
Keywords: vancomycin; therapeutic response monitoring; AUC/MIC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate which is the most appropriate parameter correlates with clinical effectiveness of vancomycin: trough drug level or AUC/MIC.

DETAILED DESCRIPTION:
Several studies have shown AUC/MIC to be the better pharmacokinetic-pharmacodynamic parameter for clinical effectiveness of vancomycin. However, the 2009 consensus guideline for vancomycin therapeutic monitoring continued to recommend trough serum concentration monitoring in the clinical setting. In 2011, Patel et al showed that highly difference between AUC(72-96h) and Cmin(96h). Different dosing and creatinine clearance may reach the same trough drug level with different AUC. The investigators wonder whether trough drug level can serve as a substitute marker for AUC and as a parameter for vancomycin therapeutic monitoring.

In this study, the investigators will calculate AUC/MIC of vancomycin with published formula, analyze its correlation with patient's clinical outcome and compare that with trough drug level.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of National Taiwan University Hospital
* Age above or equal to 20 years old
* Positive methicillin-resistant Staphylococcus aureus blood culture
* Receiving vancomycin therapy for definitive use
* Undergoing therapeutic drug monitoring (had serum vancomycin concentration level)

Exclusion Criteria:

* Age below 20 years old
* Without details of vancomycin dose and frequency
* Vancomycin treatment shorter than 72 hours
* Without renal function data (serum creatinine level, creatinine clearance)
* Without infection-related clinical outcomes (lab data such as white blood cell count , seg, C reactive protein , body temperature records)
* Receiving renal replacement therapy
* Therapeutic drug monitoring before reaching steady state
* With abnormal and undefined serum concentration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients of National Taiwan University Hospital. During the period of 2001/1/1 to 2013/12/31, age above or equal to 20 year-old adult with positive methicillin-resistant Staphylococcus aureus blood culture who receiving vancomycin therapy with therapeutic monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
30-day mortality | Day 30 after index date (the date of positive methicillin-resistant Staphylococcus aureus blood culture)

SECONDARY OUTCOMES:
90-day mortality | Day 90 after index date (the date of positive methicillin-resistant Staphylococcus aureus blood culture)
In-hospital mortality | Discharge day

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiuan Shen, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan